CLINICAL TRIAL: NCT03866213
Title: Validation of a Low-Cost, Point-of-Care Bilirubin Measurement to Diagnose Neonatal Jaundice and Monitor Phototherapy in Hospitals in Sub-Saharan Africa
Brief Title: Validation of a Jaundice Diagnostic and Monitoring Device for Low-Resource Settings
Status: Recruiting | Type: Observational
Sponsor: William Marsh Rice University (Other)
Collaborators: Kamuzu University of Health Sciences (Other); Lagos University Teaching Hospital (LUTH) (Unknown)
Responsible Party: Sponsor
Other Study IDs: BiliSpec-COMREC
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Hyperbilirubinemia, Neonatal; Jaundice, Neonatal
Keywords: Diagnostic; Point-of-Care; Low-Resource Setting
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Jaundice, Neonatal; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Quantitative Measurement of Bilirubin: Bilirubin content of the neonate will be measured by the following: BiliSpec, laboratory spectophotometric bilirubinometer (Reichert UNISTAT), and transcutaneous bilirubinometer. The infant may or may not be receiving phototherapy treatment at the time of sample measurement.
  Interventions: Diagnostic Test: BiliSpec

INTERVENTIONS:
Diagnostic Test: BiliSpec — BiliSpec will quantitatively measure the bilirubin content of a neonatal blood sample.

SUMMARY:
A team of researchers at Rice University in partnership with clinicians at Queen Elizabeth Central Hospital created BiliSpec, a low-cost battery-powered reader designed to immediately quantify serum bilirubin levels from a small drop of whole blood applied to a lateral flow strip. The simple and affordable BiliSpec system offers a faster and more cost-effective means to detect neonatal jaundice in under-resourced clinics and determine when phototherapy is needed. The goal of this study is to validate the accuracy of the BiliSpec device in measuring bilirubin levels in neonates relative to the laboratory spectrophotometric bilirubinometer and transcutaneous bilirubinometer measurements.

DETAILED DESCRIPTION:
This study will validate the accuracy of the BiliSpec device in measuring bilirubin levels in neonates relative to a laboratory spectrophotometric bilirubinometer (Reichert UNISTAT® Bilirubinometer) and transcutaneous bilirubinometer measurements.

This study will enroll up to 500 neonates at Queen Elizabeth Central Hospital and Kamuzu Central Hospital each, for a total of up to 1000 neonates, at risk for jaundice based on clinical signs and symptoms or undergoing phototherapy for treatment of jaundice. During the pilot study, 100 participants were evaluated and 147 samples total were collected. However only 7 samples collected were over 20 mg/dL. In addition to confirming the accuracy of BiliSpec in this validation study, enough samples of clinically high bilirubin concentrations (>20mg/dL) will need to be collected to ensure the device functions properly over the intended dynamic range (0-35 mg/dL). To accomplish this, data from up to 500 participants at each location will be collected.

Informed consent will be requested from the parents of all eligible babies on the ward for this study. If the guardian does not consent, the patient's bilirubin levels will be assessed using the standard of care on the ward.

During the study, the following steps will be taken:

The trained study nurse will assess the subject for clinical complications before performing the necessary heel prick blood draw.

* A transcutaneous measurement of bilirubin and a heel stick will be performed on the neonate by a trained study nurse or clinician.
* One drop of blood will be collected on the sample card and immediately used for analysis. BiliSpec will be operated by a trained nurse or trained research assistant.
* Another drop of blood, collected in a capillary tube, will be centrifuged and then measured using the laboratory spectrophotometric bilirubinometer (Reichert UNISTAT® Bilirubinometer 1310310C). The spectrophotometric bilirubinometer will be operated by trained research assistants from the Rice department of bioengineering and the University of Malawi. Bilirubin concentration values measured by the gold standard laboratory bilirubinometer will be used to guide diagnosis.

Measurements will be made at multiple time points as indicated clinically.

The neonatal bilirubin concentration in mg/dL will be determined using the BiliSpec device, the gold standard laboratory spectrophotometric bilirubinometer, and the transcutaneous bilirubinometer described in the testing procedure. Measurements of bilirubin levels will be compared. All data will be recorded using a pre-determined data collection form. Analysis of the usability and robustness of BiliSpec will also be performed with regards to usability and device function by maintaining a log of any user error in using the device and a log of any observed device malfunctions. Data will also be collected on the effectiveness of BiliSpec to monitor neonates undergoing phototherapy.

Personal identifiers will be removed and confidentiality of the subjects will be strictly preserved. The data will be kept on a secure server accessible only to the study personnel.

ELIGIBILITY:
Inclusion Criteria:

* The patient is currently being treated at Queen Elizabeth Central Hospital or Kamuzu Central Hospital in the neonatal ward.
* The patient is less than 28 days old (neonate).
* The patient is deemed to be at risk for jaundice or the patient is undergoing blue light phototherapy for treatment of jaundice.
* The patient's parent or guardian has provided informed consent for their child to participate.

Exclusion Criteria:

* Parent or guardian is unable or unwilling to provide informed consent.
* The patient is unable to receive a blood draw/heel stick as determined by their clinician.

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients currently being treated at Queen Elizabeth Central Hospital or Kamuzu Central Hospital in the neonatal ward, who are less than 28 days old (neonate), and deemed to be at risk for jaundice or the patient is undergoing blue light phototherapy for treatment of jaundice.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Device Accuracy | Total duration of hospital stay while inclusion criteria are met (<10 minutes per sample)
  Bilirubin content measured by the BiliSpec device compared against the Reichert UNISTAT laboratory spectophotometric bilirubinometer as well as a transcutaneous bilirubinometer.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Richards-Kortum, PhD, Principal Investigator — William Marsh Rice University; Maria Oden, PhD, Principal Investigator — William Marsh Rice University; Queen Dube, MD, Principal Investigator — Kamuzu University of Health Sciences; Msandeni Chiume, MD, Principal Investigator — Kamuzu University of Health Sciences
Locations (3):
- Rice University, Houston, Texas, United States
- Malawi (2):
  - Queen Elizabeth Central Hospital, Blantyre
  - Kamuzu Central Hospital, Lilongwe

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary outcome measures will be made available.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Keahey PA, Simeral ML, Schroder KJ, Bond MM, Mtenthaonnga PJ, Miros RH, Dube Q, Richards-Kortum RR. Point-of-care device to diagnose and monitor neonatal jaundice in low-resource settings. Proc Natl Acad Sci U S A. 2017 Dec 19;114(51):E10965-E10971. doi: 10.1073/pnas.1714020114. Epub 2017 Dec 4. PMID 29203650
- [Derived] Shapiro A, Anderson J, Mtenthaonga P, Kumwenda W, Bond M, Schwarz R, Carns J, Johnston R, Dube Q, Chiume M, Richards-Kortum R. Evaluation of a Point-of-Care Test for Bilirubin in Malawi. Pediatrics. 2022 Aug 1;150(2):e2021053928. doi: 10.1542/peds.2021-053928. PMID 35799070

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/13/NCT03866213/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/13/NCT03866213/ICF_001.pdf